CLINICAL TRIAL: NCT04167670
Title: A Phase 3 Randomized Multicenter Study to Evaluate the Efficacy and Safety of Open-Label Dual Therapy With Oral Vonoprazan 20 mg or Double-Blind Triple Therapy With Oral Vonoprazan 20 mg Compared to Double-Blind Triple Therapy With Oral Lansoprazole 30 mg Daily in Patients With Helicobacter Pylori Infection
Brief Title: Efficacy and Safety of Vonoprazan Compared to Lansoprazole in Participants With Helicobacter Pylori Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Phathom Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-301; 2019-002668-28 (EudraCT Number)
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Vonoprazan; Lansoprazole
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Clarithromycin; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The triple therapy arms will be blinded to participants, care providers, investigators and outcome assessors. The dual therapy arm will only blinded to the outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vonoprazan dual therapy (Experimental): Participants will receive vonoprazan 20 mg twice daily (BID) in conjunction with amoxicillin 1 g, three times daily, for 14 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- Vonoprazan triple therapy (Experimental): Participants will receive vonoprazan 20 mg twice daily (BID) in conjunction with amoxicillin 1 g BID and clarithromycin 500 mg, BID, for 14 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Clarithromycin
- Lansoprazole triple therapy (Active Comparator): Participants will receive lansoprazole 30 mg twice daily (BID) in conjunction with amoxicillin 1 g BID and clarithromycin 500 mg BID, for 14 days.
  Interventions: Drug: Amoxicillin; Drug: Clarithromycin; Drug: Lansoprazole

INTERVENTIONS:
Drug: Vonoprazan — Over-encapsulated tablets administered orally.
  Arms: Vonoprazan dual therapy; Vonoprazan triple therapy
Drug: Amoxicillin — Capsules administered orally.
Drug: Clarithromycin — Tablets administered orally.
  Arms: Lansoprazole triple therapy; Vonoprazan triple therapy
Drug: Lansoprazole — Over-encapsulated capsules administered orally.
  Arms: Lansoprazole triple therapy

SUMMARY:
To compare the efficacy of Helicobacter pylori (HP) eradication with vonoprazan dual and triple therapy regimens versus lansoprazole triple therapy regimen in participants with HP infection, excluding participants who had a clarithromycin or amoxicillin resistant strain of HP at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is ≥ 18 years of age at the time of informed consent signing.
2. In the opinion of the investigator or sub-investigators, the participant is capable of understanding and complying with protocol requirements.
3. The participant signs and dates a written, informed consent form (ICF) and any required privacy authorization prior to the initiation of any study procedures. The participant is informed of the full nature and purpose of the study, including possible risks and side-effects. The participant has the ability to cooperate with the investigator. Ample time and opportunity should be given to read and understand verbal and/or written instructions.
4. The participant has at least one of the following clinical conditions with confirmed HP+ infection demonstrated by a positive 13C-UBT during the Screening Period.

   * Dyspepsia (i.e. pain or discomfort centered in the upper abdomen) lasting at least 2 weeks
   * A confirmed diagnosis of functional dyspepsia
   * A recent / new diagnosis of (non-bleeding) peptic ulcer
   * A history of peptic ulcer not previously treated for HP infection
   * A requirement for long-term non-steroidal anti-inflammatory drug (NSAID) treatment at a stable dose of the NSAID
5. A female participant of childbearing potential who is or may be routinely sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from the signing of informed consent until Day -2 and two forms of adequate contraception from Day -1 until 4 weeks after the last dose of study drug.

Exclusion Criteria:

1. The participant has previously been treated with any regimen to attempt to eradicate HP.
2. The participant has gastric or duodenal ulcer with endoscopic evidence of current or recent bleeding.
3. The participant has confirmed diagnosis of gastric cancer by biopsy.
4. The participant is receiving colchicine.
5. The participant has received any investigational compound (including those in post marketing studies) within 30 days prior to the start of the Screening Period. A participant who has screen failed from another clinical study and who has not been dosed may be considered for enrollment in this study.
6. The participant is a study site employee, an immediate family member, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling) or who may have consented under duress.
7. The participant has cutaneous lupus erythematosus or systemic lupus erythematosus.
8. The participant has had clinically significant upper or lower gastrointestinal bleeding within 4 weeks prior to randomization.
9. The participant has Zollinger-Ellison syndrome or other gastric acid hypersecretory conditions.
10. The participant has a history of hypersensitivity or allergies to vonoprazan (including the formulation excipients: D-mannitol, microcrystalline cellulose, hydroxypropyl cellulose, fumaric acid, croscarmellose sodium, magnesium stearate, hypromellose, macrogol 8000, titanium oxide, red or yellow ferric oxide), PPIs, amoxicillin and/or clarithromycin, or any excipients used in the 13C-UBT: mannitol, citric acid or aspartame. Skin testing may be performed according to local standard practice to confirm hypersensitivity.
11. The participant has a history of alcohol abuse, illegal drug use, or drug addiction within the 12 months prior to screening, or who regularly consume >21 units of alcohol (1 unit = 12 oz/300 mL beer, 1.5 oz/25 mL hard liquor/spirits, or 5 oz/100 mL wine) per week based on self-report. Participants must have a negative urine drug screen for cannabinoids/ tetrahydrocannabinol and non-prescribed medications at screening.
12. The participant is taking any excluded medications or treatments listed in the protocol.
13. If female, the participant is pregnant, lactating, or intending to become pregnant before, during, or within 4 weeks after participating in this study; or intending to donate ova during such time period.
14. The participant has a history or clinical manifestations of significant central nervous system, cardiovascular, pulmonary, hepatic, renal, metabolic, other gastrointestinal, urological, endocrine or hematological disease that, in the opinion of the investigator, would confound the study results or compromise participants safety.
15. The participant requires hospitalization or has surgery scheduled during the course of the study or has undergone major surgical procedures within 30 days prior to the Screening Visit.
16. The participant has a history of malignancy (including MALToma) or has been treated for malignancy within 5 years prior to the start of the Screening Period (Visit 1) (the participant may be included in the study if he/she has cured cutaneous basal cell carcinoma or cervical carcinoma in situ).
17. The participant has acquired immunodeficiency syndrome or human immunodeficiency virus infection, or tests positive for the hepatitis B surface antigen, hepatitis C virus (HCV) antibody or HCV RNA. However, participants who test positive for HCV antibody, but negative for HCV RNA are permitted to participate.
18. The participant has any of the following abnormal laboratory test values at the start of the Screening Period:

    1. Creatinine levels: >2 mg/dL (>177 μmol/L).
    2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × the upper limit of normal (ULN) or total bilirubin >2 × ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1046 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Phathom Pharmaceuticals
Locations (153):
- United States (106):
  - Pinnacle Research Group, Anniston, Alabama
  - North Alabama Research Center, LLC, Athens, Alabama
  - Synexus Clinical Research US, Inc. - Alabama, Birmingham, Alabama
  - Medical Affiliated Research Center Inc, Huntsville, Alabama
  - Synexus Clinical Research US, Inc. - East Valley Family Physicians, PLC, Chandler, Arizona
  - Synexus Clinical Research US, Inc. - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Synexus Clinical Research US, Inc. - Desert Clinical Research, LLC, Mesa, Arizona
  - Elite Clinical Studies - Phoenix - BTC - PPDS, Phoenix, Arizona
  - Hope Research Institute LLC, Phoenix, Arizona
  - Del Sol Research Management - BTC - PPDS, Tucson, Arizona
  - Preferred Research Partners - ClinEdge - PPDS, Little Rock, Arkansas
  - Applied Research Center of Little Rock, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Atria Clinical Research - BTC - PPDS, North Little Rock, Arkansas
  - Anaheim Clinical Trials LLC, Anaheim, California
  - GW Research, Inc. - ClinEdge - PPDS, Chula Vista, California
  - eStudySite - Chula Vista - PPDS, Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - HB Clinical Trials, Inc., Fountain Valley, California
  - OM Research LLC - Lancaster - ClinEdge - PPDS, Lancaster, California
  - Torrance Clinical Research Institute, Lomita, California
  - Southern California Research Institute Medical Group, Inc., Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - Palmtree Clinical Research, Palm Springs, California
  - Precision Research Institute, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Paragon Rx Clinical, Inc., Santa Ana, California
  - Synexus Clinical Research US, Inc., Colorado Springs, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Riverside Clinical Research, Edgewater, Florida
  - Research Centers of America - ERG, Hollywood, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - ENCORE Borland-Groover Clinical Research - ERN - PPDS, Jacksonville, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Jesscan Medical Research, Miami, Florida
  - Nuren Medical and Research Center, Miami, Florida
  - Premier Research Associate-Miami, Miami, Florida
  - G. Medical Center, Orlando, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Synexus Clinical Research US, Inc. - St. Petersburg, Pinellas Park, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Guardian Angel Research Center, Tampa, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Nexgen Research Center, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - In Quest Medical Research - ClinEdge - PPDS, Peachtree Corners, Georgia
  - IL Gastroenterology Group, Gurnee, Illinois
  - Summit Digestive & Liver Disease Specialists, Oakbrook Terrace, Illinois
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Clinical Trials Management LLC, Covington, Louisiana
  - CroNOLA, LLC., Houma, Louisiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Meridian Clinical Research-(Rockville Maryland), Rockville, Maryland
  - Clinical Associates, Towson, Maryland
  - Oakland Medical Research Center, Troy, Michigan
  - The Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Synexus Clinical Research US, Inc. - Site 1, Henderson, Nevada
  - Synexus Clinical Research US, Inc. - Site 2, Henderson, Nevada
  - Sierra Clinical Research - ClinEdge - PPDS, Las Vegas, Nevada
  - Office - Site 1, Las Vegas, Nevada
  - Office - Site 2, Las Vegas, Nevada
  - Advanced Research Institute, Reno, Nevada
  - Drug Trials America - ClinEdge, Hartsdale, New York
  - Carolinas Research Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Peters Medical Research, LLC - ClinEdge - PPDS, High Point, North Carolina
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Synexus Clinical Research US, Inc. - Anderson, Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Rapid City Medical Center LLP, Rapid City, South Dakota
  - Multi Specialty Clinical Research, Johnson City, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - Synexus Clinical Research US, Inc. - Dallas, Dallas, Texas
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Precision Research Institute, LLC, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Digestive System Healthcare, Pasadena, Texas
  - Pearland Physicians, Pearland, Texas
  - Synexus Clinical Research US, Inc. - Plano, Plano, Texas
  - Quality Research Inc, San Antonio, Texas
  - Gastroenterology Research of San Antonio (GERSA), San Antonio, Texas
  - San Antonio Gastroenterology Associates Clinical Trials (SAGACT PLLC), San Antonio, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Synexus Clinical Research US, Inc. - Layton, Layton, Utah
  - Advanced Research Institute, Ogden, Utah
  - University of Utah Hospital- Health Sciences Center - PPDS, Salt Lake City, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Verity Research, Inc., Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Washington Gastroenterology, Bellevue, Washington
  - Harborview Medical Center, Seattle, Washington
- Bulgaria (9):
  - Multiprofile Hospital for Active Treatment Puls AD - PPDS, Blagoevgrad
  - University Multiprofile Hospital for Active Treatment, Pleven
  - Second Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia
  - Fourth Multiprofile Hospital for Active Treatment, Sofia
  - Diagnostic- Consultative Center Convex EOOD, Sofia
  - Synexus - Medical Center Synexus Sofia EOOD, Sofia
  - Synexus - Medical Centre Synexus Sofia EOOD (branch - Stara Zagora), Stara Zagora
- Czechia (5):
  - PreventaMed s.r.o., Olomouc
  - Synexus Czech s.r.o., Prague
  - MEDIC KRAL s.r.o., Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z. Oddeleni gastroenterolgie, Ústí nad Labem
  - Nemocnice Pardubickeho kraje, a.s. Orlickoustecka nemocnice, Interni oddeleni, Ústí nad Orlicí
- Hungary (7):
  - Synexus (DRS) - Synexus Magyarország Kft. Budapest, Budapest
  - Synexus Affiliate - Synexus Magyarorszag Kft. Debrecen, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Synexus (DRS) - Synexus Magyarorszag Kft. Gyula, Gyula
  - Synexus Affiliate BKS Research Kft. Hatvan, Hatvan
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Synexus (DRS) - Synexus Magyarország Kft. Zalaegerszeg, Zalaegerszeg
- Poland (17):
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Bydgoszcz
  - Gabinet Lekarski-Janusz Rudzinski, Bydgoszcz
  - Synexus - Czestochowa, Częstochowa
  - Synexus - Gdansk, Gdansk
  - Synexus - Gdynia, Gdynia
  - Synexus - Katowice, Katowice
  - Synexus Affiliate - Krakowskie Centrum Medyczne, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Ksawerów
  - Synexus - Lodz, Lodz
  - Santa Familia Centrum Badań Profilaktyki i Leczenia, Lodz
  - Synexus - Poznan, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Twoja Przychodnia - Szczecińskie Centrum Medyczne, Szczecin
  - Gastromed Specjalistyczne Centrum Gastrologii i Endoskopii, Torun
  - Synexus - Warsaw, Warsaw
  - Synexus - Wroclaw, Wroclaw
  - Melita Medical, Wroclaw
- United Kingdom (9):
  - Synexus - Wales Clinical Research Centre, Cardiff
  - Synexus - Lancashire Clinical Research Centre, Chorley
  - Synexus - Midlands Clinical Research Centre, Edgbaston
  - CPS Research, Glasgow
  - Synexus - Hexham Clinical Research Centre, Hexham
  - Synexus - Merseyside Clinical Research Centre, Liverpool
  - Synexus - Manchester Clinical Research Centre, Manchester
  - Synexus Thames Valley Clinical Research Centre, Reading
  - Synexus - North Tees Clinical Research Centre, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Megraud F, Graham DY, Howden CW, Trevino E, Weissfeld A, Hunt B, Smith N, Leifke E, Chey WD. Rates of Antimicrobial Resistance in Helicobacter pylori Isolates From Clinical Trial Patients Across the US and Europe. Am J Gastroenterol. 2023 Feb 1;118(2):269-275. doi: 10.14309/ajg.0000000000002045. Epub 2022 Sep 30. PMID 36191284
- [Derived] Chey WD, Megraud F, Laine L, Lopez LJ, Hunt BJ, Howden CW. Vonoprazan Triple and Dual Therapy for Helicobacter pylori Infection in the United States and Europe: Randomized Clinical Trial. Gastroenterology. 2022 Sep;163(3):608-619. doi: 10.1053/j.gastro.2022.05.055. Epub 2022 Jun 6. PMID 35679950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1046 participants were randomized at 103 study sites, including 71 in the United States and 32 in Europe.
Pre-assignment Details: A ^13C-urea breath test (^13C-UBT) was performed within 34 days prior to treatment to establish Helicobacter pylori (H pylori) infection status. 6 gastric mucosal biopsy specimens were collected to determine resistance of bacteria to clarithromycin, amoxicillin, and metronidazole antibiotics and to document H pylori infection.
  3385 participants were screened, 2339 of which were screen failures. 1046 participants were randomized and 1039 received at least 1 dose of the study drugs.
Groups:
- Vonoprazan Dual Therapy: Participants were administered oral doses of 20 milligrams (mg) vonoprazan tablets twice daily (BID) and oral doses of 1000 mg amoxicillin capsules 3 times daily (TID) from Day 1 to Day 14.
- Vonoprazan Triple Therapy: Participants were administered oral doses of 20 mg vonoprazan tablets BID from Day 1 to Day 14. Participants were also administered oral doses of 1000 mg amoxicillin capsules BID and 500 mg clarithromycin tablets BID from Day 1 to Day 14.
- Lansoprazole Triple Therapy: Participants were administered oral doses of 30 mg lansoprazole capsules BID from Day 1 to Day 14. Participants were also administered oral doses of 1000 mg amoxicillin capsules BID and 500 mg clarithromycin tablets BID from Day 1 to Day 14.
Period: Overall Study
Arm/Group | Vonoprazan Dual Therapy | Vonoprazan Triple Therapy | Lansoprazole Triple Therapy
Started | 349 | 349 | 348
Received Study Drugs | 348 | 346 | 345
Completed | 334 | 331 | 334
Not Completed | 15 | 18 | 14
Not completed — Pretreatment Event, Adverse Event, or Serious Adverse Event | 1 | 7 | 4
Not completed — Significant protocol deviation | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 3 | 3
Not completed — Voluntary Withdrawal | 0 | 1 | 1
Not completed — Withdrawal of Consent | 4 | 1 | 3
Not completed — Miscellaneous | 7 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Randomized Set - All participants randomly assigned to receive study drug regardless of whether or not they received a dose of study drug during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vonoprazan Dual Therapy | Vonoprazan Triple Therapy | Lansoprazole Triple Therapy | Total
Number analyzed (Participants) | 349 | 349 | 348 | 1046
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (13.47) | 50.7 (13.88) | 51.6 (13.61) | 51.4 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 226 | 216 | 652
  Male | 139 | 123 | 132 | 394
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 95 | 99 | 89 | 283
  Not Hispanic or Latino | 251 | 249 | 259 | 759
  Unknown or Not Reported | 3 | 1 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 316 | 307 | 312 | 935
  Black or African-American | 22 | 30 | 25 | 77
  Asian | 4 | 6 | 6 | 16
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Other | 4 | 1 | 3 | 8
  Unknown | 1 | 1 | 1 | 3
  Not Reported | 1 | 3 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Helicobacter Pylori (H Pylori) Eradication in Participants Without a Clarithromycin- or Amoxicillin-resistant Strain of H Pylori at Baseline
Description: H pylori eradication was determined by the ^13C-UBT test.
Time Frame: Baseline to 4 weeks after the last dose of study drugs (maximum duration of treatment was 2 weeks)
Population: Modified Intent-to-Treat Primary (MITTp) Analysis Set - All participants randomized into the study who had a H pylori infection documented by ^13C-UBT and biopsy (ie, culture or histology) at baseline and did not have a clarithromycin- or amoxicillin-resistant strain of H pylori at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Vonoprazan Dual Therapy | Vonoprazan Triple Therapy | Lansoprazole Triple Therapy
Number analyzed (Participants) | 265 | 262 | 255
percentage of participants | 78.5 | 84.7 | 78.8
Statistical Analysis 1: Comparison: Vonoprazan Dual Therapy vs Lansoprazole Triple Therapy; Noninferiority of vonoprazan dual therapy to lansoprazole triple therapy; Test type: Non-Inferiority — P-value based on a Farrington and Manning test with a noninferiority margin of 10%; p = 0.0037, Farrington and Manning test; Percentage Difference = -0.3, 95% CI 2-sided [-7.39 to 6.76] — The confidence interval of the difference in H pylori eradication rates between vonoprazan dual therapy and lansoprazole triple therapy was calculated via the Miettinen and Nurminen method
Statistical Analysis 2: Comparison: Vonoprazan Triple Therapy vs Lansoprazole Triple Therapy; Noninferiority of vonoprazan triple therapy to lansoprazole triple therapy; Test type: Non-Inferiority — P-value based on a Farrington and Manning test with a noninferiority margin of 10%; p < 0.0001, Farrington and Manning test; Percentage Difference = 5.9, 95% CI 2-sided [-0.75 to 12.62] — The confidence interval of the difference in H pylori eradication rates between vonoprazan triple therapy and lansoprazole triple therapy was calculated via the Miettinen and Nurminen method

2. Secondary Outcome: Percentage of Participants With Successful Helicobacter Pylori (H Pylori) Eradication in Participants With a Clarithromycin-resistant Strain of H Pylori at Baseline
Description: H pylori eradication was determined by the ^13C-UBT test.
Time Frame: Baseline to 4 weeks after the last dose of study drugs (maximum duration of treatment was 2 weeks)
Population: All participants randomized into the study who had H pylori infection documented by ^13C-UBT and biopsy (ie, culture or histology) at baseline and had a clarithromycin-resistant strain of H pylori at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Vonoprazan Dual Therapy | Vonoprazan Triple Therapy | Lansoprazole Triple Therapy
Number analyzed (Participants) | 56 | 73 | 72
percentage of participants | 69.6 | 65.8 | 31.9
Statistical Analysis 1: Comparison: Vonoprazan Dual Therapy vs Lansoprazole Triple Therapy; Superiority of vonoprazan dual therapy to lansoprazole triple therapy; Test type: Superiority — P-value based on a Farrington and Manning test with the null hypothesis difference ≤0 versus the alternative hypothesis difference >0; p < 0.0001, Farrington and Manning test; Percentage Difference = 37.7, 95% CI 2-sided [20.54 to 52.56] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vonoprazan Triple Therapy vs Lansoprazole Triple Therapy; Superiority of vonoprazan triple therapy to lansoprazole triple therapy; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Farrington and Manning test; Percentage Difference = 33.8, 95% CI 2-sided [17.74 to 48.12] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of All Participants With Successful Helicobacter Pylori (H Pylori) Eradication
Description: H pylori eradication was determined by the ^13C-UBT test.
Time Frame: Baseline to 4 weeks after the last dose of study drugs (maximum duration of treatment was 2 weeks)
Population: Modified Intent-to-Treat (MITT) Analysis Set - All participants randomized into the study who had H pylori infection documented by ^13C-UBT and biopsy (ie, culture or histology) at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Vonoprazan Dual Therapy | Vonoprazan Triple Therapy | Lansoprazole Triple Therapy
Number analyzed (Participants) | 324 | 338 | 330
percentage of participants | 77.2 | 80.8 | 68.5
Statistical Analysis 1: Comparison: Vonoprazan Dual Therapy vs Lansoprazole Triple Therapy; Superiority of vonoprazan dual therapy to lansoprazole triple therapy; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0063, Farrington and Manning test; Percentage Difference = 8.7, 95% CI 2-sided [1.86 to 15.44] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Vonoprazan Triple Therapy vs Lansoprazole Triple Therapy; Superiority of vonoprazan triple therapy to lansoprazole triple therapy; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0001, Farrington and Manning test; Percentage Difference = 12.3, 95% CI 2-sided [5.72 to 18.81]; The confidence interval of the difference in H pylori eradication rates between vonoprazan triple therapy and lansoprazole triple therapy was calculated via the Miettinen and Nurminen method

ADVERSE EVENTS:
Time Frame: Baseline to 4 weeks after the last dose of study drugs (maximum duration of treatment was 2 weeks)
Description: Safety Analysis Set - All participants who received at least 1 dose of study drugs.
Arm/Group | Vonoprazan Dual Therapy | Vonoprazan Triple Therapy | Lansoprazole Triple Therapy
All-Cause Mortality (participants affected / at risk) | 0/348 | 2/346 | 1/345
Serious Adverse Events (participants affected / at risk) | 5/348 | 6/346 | 3/345
Other Adverse Events (participants affected / at risk) | 20/348 | 27/346 | 48/345
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vonoprazan Dual Therapy (N=348) | Vonoprazan Triple Therapy (N=346) | Lansoprazole Triple Therapy (N=345)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vonoprazan Dual Therapy (N=348) | Vonoprazan Triple Therapy (N=346) | Lansoprazole Triple Therapy (N=345)
Diarrhoea (Gastrointestinal disorders) | 18 (18) | 14 (14) | 33 (33)
Dysgeusia (Nervous system disorders) | 2 (2) | 15 (15) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT04167670/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT04167670/SAP_001.pdf